CLINICAL TRIAL: NCT06351696
Title: The Effects of Low FODMAP Diets Accompanied With and Without Bromelain Supplement on Quality of Life, Disease Activity Index and Inflammation in Patients With Ulcerative Colitis With and Without Primary Sclerosis Cholangitis
Brief Title: The Effects of Bromelain Supplement in Patients With Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principle Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 43008563
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Ulcerative Colitis; Primary Sclerosing Cholangitis
MeSH Terms: conditions — Colitis, Ulcerative; Cholangitis, Sclerosing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Bromleine
  Interventions: Dietary Supplement: Bromlein
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bromlein — 1500 mg/day
  Arms: Intervention
Other: Placebo — Placebo (1500 mg/day)
  Arms: Placebo

SUMMARY:
In this study, patients with active mild to moderate UC with or without PSC will be randomized to receive either bromlein or placebo along with low FODMAP diet for 8 weeks.

IBDQ, SCCAIQ, CRP, TAC, TNF-a will be measured before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* active mild to moderate UC
* no other chronic disorders

Exclusion Criteria:

* changed the type and dosage of their medication in the last month
* those who have relapses that required hospitalization and change the type and dosage of medications during the intervention
* patients who do not want to continue the study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
SCCAIQ | At the 1st day and 8th week
  Simple clinical colitis activity index questionnaire (0-19, higher scores means higher symptoms)

SECONDARY OUTCOMES:
IBDQ | At the 1st day and 8th week
  IBD quality of life questionnaire (9-63, higher scores mean higher quality of life)
Serum TAC | At the 1st day and 8th week
  serum level of total anti-oxidant capacity
Serum hsCRP | At the 1st day and 8th week
  serum level of high sensitive C-reactive protein
Serum TNF-a | At the 1st day and 8th week
  serum level of tumor necrosis factor-a

CONTACTS AND LOCATIONS:
Overall Officials: Azita Hekmatdoost, MD, PhD, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Azita Hekmatdoost, Tehran, Middle East, Iran